CLINICAL TRIAL: NCT05037565
Title: Effectiveness of Partially Hydrolyzed Guar Gum in Improving Fecal Characteristics in Long Term Care Facility Residents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chan Tuen Ching, Honorary Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UW 20-521
Record Dates: First submitted 2021-08-27; First posted 2021-09-08 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Constipation
Keywords: constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): One group receive PHGG following study protocol (treatment group).
  Interventions: Dietary Supplement: Partially hydrolyzed guar gum
- Control group (No Intervention): This group will not receive PHGG

INTERVENTIONS:
Dietary Supplement: Partially hydrolyzed guar gum — Partially hydrolyzed guar gum (PHGG) is a vegetal, water soluble, non-viscous, non-gelling dietary fiber that is derived from guar gum, a water-soluble, viscous, gelling polysaccharide found in the seeds of Cyamopsis tetragonolobus. PHGG is available over the counter as a dietary supplement as fiber.
  Other Names: PHGG
  Arms: Treatment group

SUMMARY:
Partially hydrolyzed guar gum (PHGG) is a vegetal, water soluble, non-viscous, non-gelling dietary fiber that is derived from guar gum, a water-soluble, viscous, gelling polysaccharide found in the seeds of Cyamopsis tetragonolobus. PHGG is food for special medical purpose and available over-the-counter. It is as effective as lactulose treatment in relieving constipation associated abdominal pain in children. Up-to-date, there is no randomized study regarding the effectiveness of PHGG in reducing constipation in long term care facility residents, the investigator therefore would like to perform a prospective, randomized study to assess its effectiveness in long term care facility residents to improve fecal characteristics and its effect on use of laxative agents.

DETAILED DESCRIPTION:
This is a prospective, randomized, single blinded, parallel-group trial for the residents in long term care facilities covered by Community Geriatric Assessment Team of Queen Mary Hospital and Fung Yiu King Hospital. The investigator aim to recruit 52 subjects from those long term care facilities.

Subject fulfilling the inclusion criteria will be screened from the Community Geriatric Assessment Team (CGAT) of Fung Yiu King Hospital by the investigators. Study information will be explained to subject in detail and consent form (in Chinese) will be given to subject. Before commencing, subjects will be allowed to have one week to consider joining the study.

After informed consent, subjects will be randomly assigned into 2 groups. One group receive PHGG following study protocol (treatment group). Another group will be control group, no PHGG will be given. For treatment group, subjects will take 5g PHGG per day (which equals 4.2g dietary fiber) through mixing with 20ml water during treatment period. Since after mixing with PHGG, the water remains colorless and odorless, control group will also be given 20ml water by long term care facility staff as a blinding process to participant.

The study consist of two periods: a 2-week run-in period and a 4-week treatment period. During run-in period, patient's demographic characteristics will be recorded. Eligibility of patients to proceed to the treatment period will be determined, according to their baseline symptoms stool log. Stool frequency, stool characteristics (according to Bristol stool scale ranging from 1: hard stool to 7: liquid stool) and use of laxative medication will be recorded through a record diary given to subjects. During treatment period, both group of subjects need to record stool frequency, stool characteristics and use of laxative medication. Any adverse reaction will be recorded. Satisfaction of subjects towards PHGG will be assessed by questionnaire with quantification through Likert scale. Subjects will be instructed to maintain their usual daily activities including exercise, food habits, and medication consumption.

Outcome measures:

Primary outcome Fecal frequency (assessed by recording defecation times/day) Fecal characteristics (assessed by Bristol Stool Scale)

Secondary outcome Use of laxative agents per day

ELIGIBILITY:
Inclusion Criteria:

* Long term care facility residents at the age of 65 or above.
* All participants give written informed consent.
* Participants must be available to complete the study and comply with study procedures

Exclusion Criteria:

* Previous major surgery of the abdomen
* Use of PHGG in the 4 months prior to the study initiation
* Chronic constipation due to primary organic disorder of the large bowel e.g. neoplasia, post-radiation or inflammatory strictures
* On regular laxative treatment
* Patient with severe hypothyroidism
* Patients suffering from disease of the spine cord
* Subject receiving antibiotics within 3 month

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Change in Fecal characteristics (assessed by Bristol Stool Scale) from baseline at 4 weeks | Change from baseline stool characteristics at 4 weeks
  Fecal characteristics will be assessed at baseline and at 4 weeks after intervention by Bristol Stool scale. The change of stool characteristics from baseline at 4 weeks will be measured.
  Bristol stool scale range from 1 (hard stool) to 7 (liquid stool).

SECONDARY OUTCOMES:
Change in frequency of laxative use by participants per week | Change in frequency of laxative use by participant per week from baseline at 4 weeks
  Frequency of laxative use will be recorded at baseline and 4 weeks after intervention. The change in frequency of laxative use by participants will be measured.
  Frequency of laxative use will be quantified as "units per week" Senokot, lactulose and dulcolax are main laxative used by long term care facility residents.
  One unit of laxative is "7.5mg of senokot", "10ml lactulose" or "10mg of dulcolax".

CONTACTS AND LOCATIONS:
Overall Officials: Tuen Ching Chan, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital and Fung Yiu King Hospital, Hong Kong West Cluster, Hospital Authority, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giannini EG, Mansi C, Dulbecco P, Savarino V. Role of partially hydrolyzed guar gum in the treatment of irritable bowel syndrome. Nutrition. 2006 Mar;22(3):334-42. doi: 10.1016/j.nut.2005.10.003. Epub 2006 Jan 18. PMID 16413751
- [Background] Niv E, Halak A, Tiommny E, Yanai H, Strul H, Naftali T, Vaisman N. Randomized clinical study: Partially hydrolyzed guar gum (PHGG) versus placebo in the treatment of patients with irritable bowel syndrome. Nutr Metab (Lond). 2016 Feb 6;13:10. doi: 10.1186/s12986-016-0070-5. eCollection 2016. PMID 26855665
- [Background] Polymeros D, Beintaris I, Gaglia A, Karamanolis G, Papanikolaou IS, Dimitriadis G, Triantafyllou K. Partially hydrolyzed guar gum accelerates colonic transit time and improves symptoms in adults with chronic constipation. Dig Dis Sci. 2014 Sep;59(9):2207-14. doi: 10.1007/s10620-014-3135-1. Epub 2014 Apr 8. PMID 24711073
- [Background] Patrick PG, Gohman SM, Marx SC, DeLegge MH, Greenberg NA. Effect of supplements of partially hydrolyzed guar gum on the occurrence of constipation and use of laxative agents. J Am Diet Assoc. 1998 Aug;98(8):912-4. doi: 10.1016/S0002-8223(98)00210-7. No abstract available. PMID 9710664
- [Background] Yasukawa Z, Inoue R, Ozeki M, Okubo T, Takagi T, Honda A, Naito Y. Effect of Repeated Consumption of Partially Hydrolyzed Guar Gum on Fecal Characteristics and Gut Microbiota: A Randomized, Double-Blind, Placebo-Controlled, and Parallel-Group Clinical Trial. Nutrients. 2019 Sep 10;11(9):2170. doi: 10.3390/nu11092170. PMID 31509971
- [Background] Finley JW, Soto-Vaca A, Heimbach J, Rao TP, Juneja LR, Slavin J, Fahey GC. Safety assessment and caloric value of partially hydrolyzed guar gum. J Agric Food Chem. 2013 Feb 27;61(8):1756-71. doi: 10.1021/jf304910k. Epub 2013 Feb 12. PMID 23347282
- [Derived] Chan TC, Yu VMW, Luk JKH, Chu LW, Yuen JKY, Chan FHW. Effectiveness of Partially Hydrolyzed Guar Gum in Reducing Constipation in Long Term Care Facility Residents: A Randomized Single-Blinded Placebo-Controlled Trial. J Nutr Health Aging. 2022;26(3):247-251. doi: 10.1007/s12603-022-1747-2. PMID 35297467